CLINICAL TRIAL: NCT03144804
Title: A Phase 2 Study of Lamivudine in Patients With p53 Mutant Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aparna Parikh, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-044
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lamivudine; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lamivudine (Experimental): * Lamivudine administered orally every 4 weeks
  * Treatment cycles will last 28 consecutive days
  * The dosage will be determine by the PI
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Lamivudine — This drug may help prevent the growth and spread of the cancer cells to other parts of the body.
  Other Names: Combivir

SUMMARY:
This research study is studying a drug as a possible treatment for p53 mutant metastatic colorectal cancer.

The drug involved in this study is:

-Lamivudine

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved lamivudine for this specific disease but it has been approved for other uses.

In this research study, the investigators are studying the effects of lamivudine on this type of cancer. This drug may help prevent the growth and spread of the cancer cells to other parts of the body. The investigators have discovered that this particular type of colon cancer, which has a p53 mutation may be sensitive to treatment with lamivudine by impairing the ability of the cancer cells to grow.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the colon that has metastasized (stage 4) and is TP53 mutant/deleted by a CLIA approved genetic test. Only known loss of function TP53 mutation/deletion will be eligible for this study.
* Participants must have measureable disease, defined as at least on lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as > 20mm with conventional techniques or > 10 mm with spiral CT scan, MRI or calipers by clinical exam. See section 11 for evaluation of measurable disease
* Patients must be resistant to or intolerant of 5FU, oxaliplatin, irinotecan, bevacizumab and cetuximab/panitumumab (if RAS wild type)
* Age 18 or older.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 8 weeks.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,200/mcL
  * platelets ≥75,000/mcL
  * total bilirubin ≤1.5 × institutional upper limit of normal within normal
  * AST(SGOT)/ALT(SGPT) ≤5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of lamivudine on the developing human fetus are known to be teratogenic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of lamivudine administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lamivudine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because lamivudine is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lamivudine, breastfeeding should be discontinued if the mother is treated with lamivudine.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lamivudine
* HBV positive participants will be excluded given the known effects of lamivudine on HBV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna R. Parikh, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts general Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamivudine: * Lamivudine administered orally every 4 weeks
  * Treatment cycles will last 28 consecutive days
  * The dosage will be determine by the PI
  Lamivudine: This drug may help prevent the growth and spread of the cancer cells to other parts of the body.
Period: Overall Study
Arm/Group | Lamivudine
Started | 36
Completed | 32
Not Completed | 4
Not completed — 4 participants had disease progression within 1 month of study treatment and were deemed unevaluable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lamivudine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan or MRI, complete response (CR) is the disappearance of all target lesions and partial response (PR) is a >/=30% decrease in the sum of the longest diameter of target lesions. Overall Response (OR) = CR + PR. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Lamivudine
Number analyzed (Participants) | 32
participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Time Frame: 2 years
Population: Of the 32 analyzed participants, 5 participants were censored in PFS analysis because they were taken off treatment before their first radiographic progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lamivudine
Number analyzed (Participants) | 27
days | 56 [55 to 92]

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lamivudine
Number analyzed (Participants) | 36
days | 186 [129 to 276]

4. Secondary Outcome: Overall Disease Control Rate
Description: Disease control rate (DCR) describes the percentage of patients with advanced cancer whose therapeutic intervention has led to a complete response (CR), partial response (PR), or stable disease (SD) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria:
  * CR is the disappearance of all target lesions
  * PR is at least a 30% decrease in the sum of the longest diameters of target lesions
  * SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD)
  * PD is at least a 20% increase in the sum of the longest diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lamivudine
Number analyzed (Participants) | 36
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of protocol therapy up until participants were taken off study, a median of approximately 7 months.
Description: Adverse events were evaluated through regular investigator assessment and regular laboratory testing.
Arm/Group | Lamivudine
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 9/36
Other Adverse Events (participants affected / at risk) | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamivudine (N=36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Death NOS (General disorders) | 1 (1)
Vaginal bleeding (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1) — Central chest pain with deep inspiration
Fatigue (General disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Osteomyelitis (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) — small bowel obstruction
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lamivudine (N=36)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 14 (19)
Alanine aminotransferase increased (Investigations) | 5 (10)
Alkaline phosphatase increased (Investigations) | 17 (24)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 19 (50)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Anxiety (Psychiatric disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 13 (20)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 7 (11)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Chills (General disorders) | 3 (5)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Creatinine increased (Investigations) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Dizziness (Nervous system disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 20 (22)
Fever (General disorders) | 6 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Loose stools
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Intermittent melena
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Indigestion
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (53)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (11)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 14 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (9)
Hypothermia (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations - Other (Investigations) | 1 (1) — Reduced Plasma Bicarbonate
Irritability (General disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 18 (54)
Malaise (General disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (19)
Neutrophil count decreased (Investigations) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Palpitations (Cardiac disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Platelet count decreased (Investigations) | 5 (9)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Skin/subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Skin irritation
Skin/subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Perirectal irritation
Urinary tract infection (Infections and infestations) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (10)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 7 (13)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Vaginal bleeding
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Central chest pain with deep inspiration
General disorders and administration site conditions - Other (General disorders) | 1 (1) — occasional mild sweats
General disorders and administration site conditions - Other (General disorders) | 1 (1) — night sweats
General disorders and administration site conditions - Other (General disorders) | 1 (1) — sore on left inner cheek
General disorders and administration site conditions - Other (General disorders) | 1 (1) — water ostomy
General disorders and administration site conditions - Other (General disorders) | 1 (1) — numbness on chest
General disorders and administration site conditions - Other (General disorders) | 1 (1) — new lump on breast
General disorders and administration site conditions - Other (General disorders) | 1 (1) — weakness
General disorders and administration site conditions - Other (General disorders) | 1 (1) — blood in stool
General disorders and administration site conditions - Other (General disorders) | 1 (1) — hepatomegaly
General disorders and administration site conditions - Other (General disorders) | 1 (1) — leg cramps
General disorders and administration site conditions - Other (General disorders) | 1 (1) — rash unspecified
General disorders and administration site conditions - Other (General disorders) | 1 (1) — development of right inguinal hernia
General disorders and administration site conditions - Other (General disorders) | 1 (1) — numbness
General disorders and administration site conditions - Other (General disorders) | 1 (1) — inflammation
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — intermittent abdominal discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03144804/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03144804/ICF_001.pdf